CLINICAL TRIAL: NCT00124033
Title: Management of CBD Stones at Laparoscopic Cholecystectomy: A NSW Collaborative Prospective Randomised Trial to Assess the Value of Transcystically Inserted CBD Stents to Facilitate Post-Operative ERCP
Brief Title: Management of Common Bile Duct (CBD) Stones at Laparoscopic Cholecystectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: South West Sydney Local Health District (Other)
Collaborators: Catholic Health Care Services (Other); Greater Western Area Health Service (Unknown); Hunter New England Area Health Service (Unknown); Northern Sydney and Central Coast Area Health Service (Other); South Eastern Area Health Service (Other); Sydney South West Area Health Service (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 04/001
Record Dates: First submitted 2005-07-25; First posted 2005-07-26 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2005-06

CONDITIONS: Choledocholithiasis; Cholelithiasis
Keywords: Cholecystectomy; Cholangiopancreatography, Endoscopic Retrograde
MeSH Terms: conditions — Choledocholithiasis; Cholelithiasis

INTERVENTIONS:
Procedure: Transcystic Stenting (Facilitated ERCP)

SUMMARY:
This study is designed to assess whether a new technique called facilitated endoscopic retrograde cholangiopancreatography (ERCP) is or is not superior to conventional ERCP for removing stones found in the bile duct at the time of laparoscopic cholecystectomy. ERCP is an endoscopic procedure used to facilitate the radiological examination and subsequent manipulation of the common bile duct (eg. opening it up, which is called sphincterotomy). Both facilitated and conventional ERCP are performed as a separate procedure after the initial gallbladder surgery. This is a comparative study of these two techniques in a randomised clinical trial.

The aim of this randomised clinical trial is to enable surgeons to decide whether placement of a plastic stent at the time of laparoscopic cholecystectomy will improve the success rate and safety of subsequent ERCP and sphincterotomy.

DETAILED DESCRIPTION:
Symptomatic gallstone disease is common. In the year July 2001-2002, laparoscopic cholecystectomy was performed on 5,235 patients in NSW public hospitals. Up to 18% of patients undergoing laparoscopic cholecystectomy for gallstones may have concomitant common bile duct stones (choledocholithiasis). Twenty-five percent of bile duct stones are completely unsuspected. Therefore the optimal management of bile duct stones is a significant issue for all general surgeons who perform this very common operation. Yet, the management of these patients in the laparoscopic era remains contentious.

Prior to the laparoscopic era cholecystectomy patients with bile duct stones were managed surgically during open cholecystectomy (OC), with direct exploration of their common bile duct (choledochotomy). However, open surgical bile duct exploration waned in popularity and progressively stones were dealt with endoscopically, either pre or post cholecystectomy. As laparoscopic technology advances, simultaneous clearance of the bile duct at the time of laparoscopic cholecystectomy is regaining popularity.

Some surgeons elect to remove bile duct stones at the index operation through the cystic duct. This approach has a success rate of between 75 and 90%. When there is failure to clear the bile duct transcystically, some surgeons proceed to a choledochotomy to clear the duct, while others close the cystic duct stump, leaving the stones in situ to be removed at a later date by endoscopic retrograde cholangiopancreatography (ERCP) and sphincterotomy. The argument in favour of immediate choledochotomy is that the duct may be cleared in one sitting. The argument against it is that the morbidity of choledochotomy is considerable. The argument for a subsequent ERCP is that the morbidity of choledochotomy is avoided. The argument against subsequent ERCP is that there may be difficulty cannulating the common bile duct and that ERCP with sphincterotomy is associated with a significant morbidity, particularly pancreatitis.

An alternative approach taken by the majority of surgeons in NSW when confronted by common bile duct stones at laparoscopic cholecystectomy is to close the cystic duct stump in all patients, without exploring the duct transcystically. Stones are left in situ, to be removed at a later date endoscopically - by ERCP and sphincterotomy. The attendant risks of this approach are mentioned above.

Another approach is to facilitate the performance of post-operative ERCP and sphincterotomy by inserting a stent transcystically at the time of laparoscopic cholecystectomy. Facilitated ERCP has recently been reported in a prospective consecutive series from Nepean Hospital. Failure to access the common bile duct at first attempt was 1.2% in this series, which compares favourably with duct access failure rates - reported in the literature - of 5-12% without the facilitation of a stent. The incidence of pancreatitis, bleeding and duodenal perforation after facilitated ERCP was 0%, 0% and 0.6%, respectively. Two cases (1.2%) of cholangitis were also reported. Comparison to other series suggests that facilitated ERCP offers real advantages over the conventional unfacilitated ERCP for bile duct stone removal, which has a reported pancreatitis rate of 2-11% (and our own rate of 8%); a bleeding rate of 2-4 % and a duodenal perforation rate of 1-4%. The mortality rates of these ERCP techniques cannot be compared at this preliminary stage because of insufficient numbers in the Nepean series.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be able to give informed consent preoperatively (i.e. elective procedures only)
* Patients at higher than normal risk of having CBD stones identified at OC. For example: *CBD stones identified at ultrasound; *Wide CBD (>6mm) at ultrasound; *Previous, recent, current cholangitis, jaundice, or biliary pancreatitis; or *Abnormal AST and ALT levels (>2 times normal).

Exclusion Criteria:

* Pregnancy at time of surgery
* Patients not fit for surgery. For example: *Those with acute cholecystitis or persistent obstructive jaundice; *Patients who have had a previous ERCP and sphincterotomy; or *Patients in whom intervention was not technically possible (eg. previous Billroth II gastrectomy).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340
Dates: Start 2004-03; Study Completion 2015-12

PRIMARY OUTCOMES:
Safety of facilitated ERCP compared to conventional unfacilitated ERCP - as assessed by the incidence of pancreatitis post ERCP

SECONDARY OUTCOMES:
The success rate and morbidity of transcystic exploration for common bile duct stone removal across a broad spectrum of surgeons
The success rate of transcystic stent placement across a broad spectrum of surgeons
The overall morbidity of post-operative ERCP, with further comparisons of the morbidity of facilitated and conventional ERCP, with and without transcystic exploration of the common bile duct to remove stones
Hospitalisation time according to treatment group
The incidence of hyperamylasemia after transcystic exploration of the common bile duct, transcystic insertion of a stent or transcystic cholangiography alone
The success rate and complications after choledochotomy for common bile duct stones
The failure rate of selective common bile duct cannulation for facilitated ERCP as compared to conventional ERCP
Incidence of multiple endoscopic procedures when the common bile duct was not explored at the primary operation and whether or not this is affected by facilitation at ERCP
Long-term efficacy of techniques used to remove common bile duct stones, as measured by the recurrence of stones in the bile duct

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Martin, MBBS MSc, Principal Investigator — Sydney West Area Health Service (Department of Surgery, Nepean Hospital)
Locations (13):
- Australia (13):
  - Bankstown-Lidcombe Hospital, Bankstown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Dubbo Base Hospital, Dubbo, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Blue Mountains District ANZAC Memorial Hospital, Katoomba, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Hawkesbury District Health Service, Windsor, New South Wales

REFERENCES:
- [Background] Martin CJ, Cox MR, Vaccaro L. Laparoscopic transcystic bile duct stenting in the management of common bile duct stones. ANZ J Surg. 2002 Apr;72(4):258-64. doi: 10.1046/j.1445-2197.2002.02368.x. PMID 11982511